CLINICAL TRIAL: NCT00872443
Title: Interest of Occlusion of Permeable Foramen Ovale After a Cryptogenic Cerebrovacular Accident.
Brief Title: Interest of Occlusion of Permeable Foramen Ovale After a Cryptogenic Cerebrovascular Accident (CVA)
Acronym: FOPasa
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Dr Patrice Guerin, Nantes University Hospital
Other Study IDs: BRD 08/8-J
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Permeable Foramen Ovale; Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FOP: Patients who already have an occlusion of POF secondary to a cryptogenic CVA and younger than 55 years old and without characterized thromboembolic events.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Collection of characteristics of interauricular septum, characteristics of the CVA, and headache history.
  Collection of anamnesis data, surgical past history, especially at the moment of the implement of prothesis, collection of dtat of transthoracic echography, transcranial echodoppler, holter ECG, cerebral MRI.

SUMMARY:
Facing the lack of recommandations of Neurology and cardiology societies, the investigators decided in 2002 some Good Medical Practices to define a specific and precise population for whom the closure of permeable oval formaen after a first CVA seem to be necessary. Current survey of these patients after implantation of a prothesis in interauricular septum is defined by a consultation at 1, 3 and 6 months after surgery for a clinical exam and an echocardiography. One year after implantation, the investigators systematically realized a control by MRI associated to a contrast echography.

In the aim of evaluating the investigators' medical practice, the investigators decided to do an observational study which will permit us to judge of the interest or lack of interest of our "Good medical practice" before the publication of prospective and randomised clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* less than 55 years old
* occlusion of FOP after cryptogenic CVA

Exclusion Criteria:

* characterized thromboembolic event
* patients who have a surgery after transitory ischemic accident

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patient who had an occlusion of POF after CVA, younger than 55 years and without thromboembolic events.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France